CLINICAL TRIAL: NCT05214924
Title: Assessment of the Effectiveness of Intra-articular Injectable Platelet-rich Fibrin (iPRF) Injections in the Management of Mild and Moderate Degeneration of the Temporomandibular Joints
Brief Title: Effectiveness of iPRF Injections in Temporomandibular Joints Degeneration Management
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Joanna Smardz, Investigator, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMU2/2021
Record Dates: First submitted 2021-12-27; First posted 2022-01-31 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Disorder; Temporomandibular Joint Disorders; Temporomandibular Arthritis; Temporomandibular Joint Osteoarthritis
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injectable platelet-rich fibrin injection (Experimental): Each of the participants from iPRF injection group will receive two injections of iPRF with an interval of 30 days.
  Interventions: Biological: Injectable platelet-rich fibrin
- Platelet-rich plasma injection (Active Comparator): Each of the participants from PRP injection group will receive two injections of PRP with an interval of 30 days.
  Interventions: Biological: Platelet-rich plasma

INTERVENTIONS:
Biological: Injectable platelet-rich fibrin — Intra-articular injection of injectable platelet-rich fibrin into temporomandibular joint/joints with diagnosed mild to moderate degenerative joint disease.
  Other Names: iPRF
  Arms: Injectable platelet-rich fibrin injection
Biological: Platelet-rich plasma — Intra-articular injection of platelet-rich plasma into temporomandibular joint/joints with diagnosed mild to moderate degenerative joint disease.
  Other Names: PRP
  Arms: Platelet-rich plasma injection

SUMMARY:
The aim of the study is to evaluate the effectiveness of intra-articular platelet-rich fibrin (iPRF) injections in the management of moderate and mild cases of degeneration of the temporomandibular joints. This randomized, two-arm controlled trial will involve 42 adult patients diagnosed with mild or moderate degeneration of the temporomandibular joints on the basis of clinical examination and magnetic resonance imaging or computed tomography. Qualified study participants will be randomly assigned to two groups. The studied group will receive two injections of iPRF with an interval of 30 days, while the control group will receive injections of platelet-rich plasma (PRP) during this time. Each subject will be tested on the day of the first injection (D0), on the day of the second injection (D30), and then 60 (D60) and 12 (D120) days after the first injection using MRI/CT, Doppler Hi-dop, clinical examination and surveys.

DETAILED DESCRIPTION:
Background: The term temporomandibular disorders is used to describe a wide spectrum of functional modifications and pathological conditions involving the temporomandibular joints, masticatory muscles and other surrounding structures. Temporomandibular disorders are the second most common cause of pain symptoms in the craniofacial area. It is estimated that they may affect up to 56% of the adult Polish population. One of the most common forms of temporomandibular disorders are intra-articular abnormalities. They can lead to degeneration within the articular surfaces and articular disc of the joints. The treatment of degeneration of the temporomandibular joints is a great therapeutic challenge. There are scientific reports suggesting that one of the effective methods may be intra-articular injections. Injectable platelet-rich fibrin (iPRF) is an autologous material obtained from human blood, which contains a high concentration of inactivated platelets, white blood cells and mesenchymal stem cells. After injection into the tissues, it initiates natural repair processes. Despite the fairly wide possibilities of application, this method has not yet been tested in terms of its use in the treatment of degeneration of the temporomandibular joints.

Aim: The aim of the study is to evaluate the effectiveness of intra-articular platelet-rich fibrin injections in the management of moderate and mild cases of degeneration of the temporomandibular joints.

Material and methods: A randomized, two-arm controlled trial will involve 42 adult patients diagnosed with mild or moderate degeneration of the temporomandibular joints on the basis of clinical examination and magnetic resonance imaging or computed tomography. Criteria for exclusion from the study will include: severe hematologic and/or neurological disorder; rheumatoid arthritis; septic arthritis; polymyalgia rheumatica; gout; Paget's disease; osteonecrosis; connective tissue disease; malignant disease; vasculitis; any previous temporomandibular joint invasive treatment; any current temporomandibular joint conservative or invasive treatment; patients who had used oral, parenteral or intra-articular corticosteroids in the 3 months prior to the first injection; previous or current radiotherapy of head and neck; pregnancy or lactation; presence of severe mental disorders; drug and/or alcohol addiction; presence of local contraindications for injection therapy; patients with needle phobia; presence of hypersensitivity to substances to be used in the study.

Qualified study participants will be randomly assigned to two groups. The studied group will receive two injections of iPRF with an interval of 30 days, while the control group will receive injections of platelet-rich plasma (PRP) during this time. The use of PRP has been already described in the scientific literature as being effective in the treatment of joint degeneration. Each subject will be tested on the day of the first injection (D0), on the day of the second injection (D30), and then 60 (D60) and 12 (D120) days after the first injection using the following methods:

1. Magnetic resonance imaging of the temporomandibular joints (D0)
2. Examination with the Doppler Hi-dop (D0, D30, D60, D120)
3. Examination of the mandibular mobility ranges with a professional ruler (D0, D30, D60, D120)
4. Clinical examination according to diagnostic criteria for temporomandibular disorders - DC / TMD International Examination Form (D0, D120)
5. Surveys: Short Form 36 (SF-36), General Oral Health Assessment Index (GOHAI (HRQoL)) (D0, D60, D120), Jaw Functional Limitation Scale-20 (D0, D30, D60, D120), TMD Pain Screener (D0, D30, D60, D120) Pain Numerical Rating Scale (D0, D30, D60, D120), Graded Chronic Pain Scale (DO, D30, D60, D120).

The collected data will then be subjected to statistical analysis in order to verify the research hypothesis and capture statistically significant relationships.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years old
* mild to moderate degenerative temporomandibular joint disease based on DC/TMD protocol and MRI/CT
* agreement to take part in the study

Exclusion Criteria:

* severe hematologic and/or neurological disorder
* rheumatoid arthritis
* septic arthritis
* polymyalgia rheumatica
* gout
* Paget's disease
* osteonecrosis
* connective tissue disease
* malignant disease
* vasculitis
* any previous temporomandibular joint (TMJ) invasive treatment
* any current temporomandibular joint (TMJ) conservative or invasive treatment
* patients who had used oral, parenteral or intra-articular corticosteroids in the 3 months prior to the first injection
* previous or current radiotherapy of head and neck
* pregnancy or lactation
* presence of severe mental disorders
* drug and/or alcohol addiction
* presence of local contraindications for injection therapy
* patients with needle phobia
* presence of hypersensitivity to substances to be used in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of intra-articular platelet-rich fibrin (iPRF) injections on TMD symptoms reduction assessed by clinical examination in accordance to Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) protocol with DC/TMD examination form. | Up to 3 months
  Each patient will undergo DC/TMD protocol-based clinical examination before and after injections using DC/TMD examination form assessing incidence of pain and disfunction in temporomandibular joints, masticatory muscles and surrounding structures.

SECONDARY OUTCOMES:
The effectiveness of intra-articular platelet-rich fibrin (iPRF) injections on the jaw mobility assessed by jaw mobility measurement with professional ruler (millimeters). | Up to 3 months
  Each participant will undergo jaw mobility assessment (measured with millimeters) with the use of professional ruler before and after injections.
The influence of intra-articular platelet-rich fibrin (iPRF) injections on intra-articular sounds assessed using Doppler Hi-dop (Hz). | Up to 3 months
  Each participant will undergo Doppler Hi-dop examination (measured in Hz) before and after injections.
The influence of intra-articular platelet-rich fibrin (iPRF) injections on pain in temporomandibular area assessed using Graded Chronic Pain Scale. | Up to 3 months
  Each participant will fill in Graded Chronic Pain Scale before and after injections. Scoring Criteria for Grading Chronic Pain Severity: Characteristic Pain Intensity is a 0 to 100 score derived from Questions 1 through 3:Mean (Pain Right Now, Worst Pain, Average Pain) X 10. Disability Score is 0 to 100score derived from Questions 4 through 6:Mean (Daily Activities, Social Activities, Work Activities) X 10. Disability Points: Add the indicated points for Disability Days (Question 7)and for Disability Score. Classification: GRADE 0- No TMD pain in prior 6 months. GRADE I-Low Intensity Characteristic Pain Intensity<50, Low Disability<3 Disability Point. GRADE II -High Intensity Characteristic Pain Intensity >50, LowDisability<3 Disability Points. GRADE III- High Disability3 to 4 Disability Points, Moderately Limiting (Regardless of Characteristic Pain Intensity). GRADE IV- High Disability 5 to 6 Disability Points, Severely Limiting (Regardless of Characteristic Pain Intensity).
The influence of intra-articular platelet-rich fibrin (iPRF) injections on reduction of pain in temporomandibular area assessed using TMD pain screener questionnaire. | Up to 3 months
  Each participant will fill in TMD pain screener questionnaire before and after injections. The first item has scores of 0-2 (a=0, b=1, c=2), while the remaining items are scored simply as a=0, b=1. A sum is computed. Higher scores mean more intense pain.
The influence of intra-articular platelet-rich fibrin (iPRF) injections on reduction of pain in temporomandibular joints assessed using Pain Numerical Rating Scale. | Up to 3 months
  Each participant will be asked to assess the pain during temporomandibular joints palpation using Pain Numerical Rating Scale before and after injections. It is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
The influence of intra-articular platelet-rich fibrin (iPRF) injections on jaw functionality assessed using Jaw Functional Limitation Scale-20. | Up to 3 months
  Each participant will fill in Jaw Functional Limitation Scale-20 before and after injections. It is organ-specific instrument comprising 3 constructs for assessing functional status of the masticatory system; the 3 scales exhibit properties that are ideal for both research and patient evaluation in patient groups with a range of functional limitations of the jaw.
The influence of intra-articular platelet-rich fibrin (iPRF) injections on quality of life using GOHAI questionnaire. | Up to 3 months
  Each participant will fill in GOHAI questionnaire before and after injections. The GOHAI assesses self-perceived oral health through 12 questions that explore the pain, discomfort, dysfunctions and the psychosocial impacts of dental diseases.
The influence of intra-articular platelet-rich fibrin (iPRF) injections on quality of life using Short Form 36 questionnaire. | Up to 3 months
  Each participant will fill in Short Form 36 (SF-36) questionnaire before and after injections. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Mieszko Wieckiewicz, Prof., Study Chair — Wroclaw Medical University
Locations (1):
- Wroclaw Medical University, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: No